CLINICAL TRIAL: NCT03046147
Title: Bone Mineral Density and Markers of Bone Turnover After Roux-en-Y Gastric Bypass
Brief Title: The Effect of Roux-en-Y Gastric Bypass on Bone Turnover
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, MD, PhD, Hvidovre University Hospital
Other Study IDs: KBM-IS-Bone
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Gastric Bypass Surgery; Obesity; Bone Loss
MeSH Terms: conditions — Obesity; Bone Diseases, Metabolic | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RYGB patients with preoperative type diabetes: Recruited from a previously investigated cohort (NCT 01202526)
  Interventions: Procedure: Roux-en-Y gastric bypass
- RYGB patients with preoperative normal glucose tolerance: Recruited from a previously investigated cohort (NCT 01202526)
  Interventions: Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — Roux-en-Y gastric bypass surgery for morbid obesity

SUMMARY:
Bone mineral density (BMD) is decreased after Roux-en-Y gastric bypass (RYGB) but whether RYGB induces changes in BMD beyond adaptation to major weight loss is not known. We aim to investigate BMD changes in weight bearing (hip, lumbal columna) and in non-weight bearing (forearm) regions before and after maximal weight loss at 1 year and after weight stabilisation at 4 years after RYGB. Moreover, plasma markers of bone turnover will be studied at fasting and during oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Participation in previos study ((NCT 01202526)

Exclusion Criteria:

* Treatment of osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a previously investigated cohort of 20 subjects undergoing Roux-en-Y gastric bypass surgery (NCT 01202526). The previous study aimed at investigating acute and long term changes in insulin sensitivity and secretion, whereas the present follow-up study investigates changes in bone metabolism as the primary outcome.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Changes in bone mineral density of non-weight bearing bone | 1 year, 4 years
  DXA scans of forearm
Changes in bone mineral density of weightbearing bone | 1 year, 4 years
  DXA scans of hip and lumbal columna

SECONDARY OUTCOMES:
Plasma markers of bone turnover | 1 week, 3 months, 1 year, 4 years
  At fasting
Plasma markers of bone turnover | 3 months, 1 year, 4 years
  during OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University hospital Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No